CLINICAL TRIAL: NCT00340431
Title: Phase 1 Study of the Safety and Immunogenicity of MSP1(42)-FVO/Alhydrogel and MSP1(42)-3D7/Alhydrogel, Asexual Blood-Stage Vaccines for Plasmodium Falciparum Malaria
Brief Title: Experimental Vaccine for Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999904216; 04-I-N216
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-02-06

CONDITIONS: Plasmodium Falciparum Malaria; Vaccines
Keywords: Human; Clinical Trial; Mosquito
MeSH Terms: conditions — Malaria, Falciparum

INTERVENTIONS:
Drug: MSP1(42)-FVO & MSP1(42)-3D7

SUMMARY:
This study will evaluate the safety of two experimental malaria vaccines in healthy volunteers and examine their immune response to them. Safety will be assessed by comparing vaccine side effects in groups of volunteers who receive increasing doses of the same vaccine (dose-escalating study). Immune response will be evaluated by comparing the levels of antibody production with each dose. (Antibodies are infection-fighting proteins produced by the immune system.) The two vaccines in this study contain different types of a malaria protein called MSP1: one type is MSP142FVO and the other is MSP1423D7.

Malaria parasites are spread from person to person by mosquitoes. There are four types of malaria parasites. The vaccine tested in this study is designed to work against Plasmodium falciparum, the parasite responsible for most deaths in children due to malaria in sub-Saharan Africa. The vaccine stimulates the body to produce antibodies that prevent P. falciparum from entering the person's red blood cells.

Healthy normal volunteers between 18 and 50 years of age may be eligible for this 12-month study, conducted at Quintiles Phase 1 Services in Lenexa, Kansas. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants receive three doses of the vaccine-on the first day of the study (day 0), at 1 month (day 28), and at 6 months (day 180) -through injection into an arm muscle. The first group of subjects receives 5 micrograms of vaccine, the second group receives 20 micrograms, and the third group receives 80 micrograms. All participants are observed in the clinic for 30 minutes after each immunization for immediate reactions to the vaccine and keep a record of their temperature and of any reactions and side effects they experience for 6 days after the vaccination. At various intervals throughout the study, participants undergo a brief physical examination and blood tests. Women of childbearing potential have a urine pregnancy test on the day of each injection.

DETAILED DESCRIPTION:
The purpose of this Phase 1 clinical trial is to evaluate the safety and immunogenicity of two asexual blood stage vaccines for Plasmodium falciparum malaria, MSP1(42)-FVO/Alhydrogel and MSP1(42)-3D7/Alhydrogel, in healthy adult volunteers. Between 2-3 million deaths occur each year as a result of malaria. Most of these deaths are a result of P. falciparum malaria, in children under five years of age, in sub-Saharan Africa. A safe and effective vaccine that would reduce both morbidity and mortality secondary to P. falciparum infection would be a valuable resource in the fight against this disease. The merozoite surface protein 1 (MSP1) is the first protein to be identified on the surface of the blood stage parasite. A portion of MSP1 is carried into the newly invaded erythrocyte on the surface of the parasite. Clinical symptoms of malaria in humans are due to the asexual blood stage. Therefore, this vaccine was designed to protect an individual from illness due to the asexual stage of P. falciparum infection by inhibiting parasite invasion of erythrocytes. The MSP1(42)/Alhydrogel vaccines have been used in five preclinical animal trials and no clinically significant risks have been identified. The study will be conducted at Quintiles Phase I Services (Lenexa, KS). We will evaluate three dose levels of both the MSP1(42)-FVO/Alhydrogel and the MSP1(42)-3D7/Alhydrogel vaccines (5 micro g, 20 micro g, 80 micro g). Sixty healthy male and non-pregnant female volunteers ages 18 to 50 will be enrolled. Ten volunteers in each group will receive a 5 micro g, 20 micro g, or 80 mirco g dose of either MSP1(42)-FVO or MSP1(42)-3D7 vaccines by intramuscular injection in an open label study on months 0, 1, and 6. The groups will be staggered such that adequate safety evaluation can be performed prior to dose escalation. The duration of the study is 12 months per volunteer. The primary objective of this trial is to determine the frequency and severity of vaccine-related adverse events for each dose. The secondary objective is to determine the dose that generates the highest serum antibody levels to homologous MSP1(42) antigen at Day 42.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females between 18 and 50 years, inclusive.

Good general health as determined by means of the screening procedure.

Available for the duration of the trial (52 weeks).

Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

Pregnancy as determined by a positive urine human chorionic gonadotrophin (Beta-hCG), if female.

Participant unwilling to use reliable contraception methods for the duration of the trial.

Currently lactating and breast-feeding (if female).

Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Evidence of obesity; BMI must be less than 35. Body mass index equals ((weight in pounds)/(height in inches) x (height in inches)) x 703.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.

Laboratory evidence of liver disease (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory).

Laboratory evidence of hematologic disease (absolute neutrophil count less than 1,5000/mm(3); hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by sex; or platelet count less than 140,000/mm(3)).

Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.

Volunteer has abused alcohol or illicit drugs during the past 6 months, by history and/or positive urine drug screen (any detectable levels) on Study Day 0 or 180.

History of a severe allergic reaction or anaphylaxis.

Severe asthma (emergency room visit or hospitalization within the last 6 months).

Positive ELISA and confirmatory Western blot tests for HIV-1.

Positive ELISA and confirmatory immunoblot tests for HCV.

Positive HBsAg by ELISA.

Known immunodeficiency syndrome.

Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or while the study is ongoing.

Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.

History of a surgical splenectomy and/or abnormal splenic function.

Receipt of blood products within the past 6 months.

Previous receipt of an investigational malaria vaccine.

Receipt of antimalarial prophylaxis during the past 12 months.

Prior malaria infection.

Travel to a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.

History of a known allergy to nickel.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0
Dates: Start 2004-06-09; Study Completion 2008-02-06

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase 1 Services, Lenexa, Kansas, United States

REFERENCES:
- [Background] McBride JS, Heidrich HG. Fragments of the polymorphic Mr 185,000 glycoprotein from the surface of isolated Plasmodium falciparum merozoites form an antigenic complex. Mol Biochem Parasitol. 1987 Feb;23(1):71-84. doi: 10.1016/0166-6851(87)90189-7. PMID 2437453